CLINICAL TRIAL: NCT06090708
Title: Effect of Mothers' Application of Yogurt Probiotic Bacteria on Relieving Their Young Children's Acute Gastroenteritis
Brief Title: Yogurt Probiotic Bacteria on Relieving Young Children Acute Gastroenteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro
Record Dates: First submitted 2023-10-09; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Acute Gastroenteritis
Keywords: Yogurt Probiotic Bacteria; young Children; Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Children with acute gastroenteritis received standard hospital care and the prescribed medication of control group for acute gastroenteritis.
- Probiotic Study Group (Experimental): Children with acute gastroenteritis received fresh probiotic yogurt (1st day of production) for three consecutive days in addition to standard hospital care and prescribed medication for acute gastroenteritis.
  Interventions: Dietary Supplement: yogurt with probiotic bacteria

INTERVENTIONS:
Dietary Supplement: yogurt with probiotic bacteria — Children in probiotic study group were received 15 mg/kg of market available fresh probiotic yogurt after stopping vomiting every four to six hours for three consecutive days beside to the standard hospital care and the prescribed medication for acute gastroenteritis.
  Arms: Probiotic Study Group

SUMMARY:
The goal of this clinical trial is to test the effect of mothers' application of yogurt probiotic bacteria on relieving their young children's acute gastroenteritis in children had two to five years old. The main hypothesis is children with acute gastroenteritis who receive yogurt probiotic bacteria exhibit less diarrhea, vomiting and dehydration than those who don't.The study subjects were divided into two equal groups (probiotic study group and control group).

ELIGIBILITY:
Inclusion Criteria:

* newly admitted children with no or some dehydration and with acute gastroenteritis.

Exclusion Criteria:

* bloody watery diarrhea

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Experience of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  yes/no
Consistency of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Soft/ watery/ abnormal constitute
Amount of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Small / moderate/ large/ severe
Frequency of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  times /day.
Odor of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  No odor/ offensive odor
Duration of diarrhea | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  /days.
Experience of Vomiting | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Yes/ no
Amount of Vomiting | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Small / moderate/ large/ severe
Frequency of Vomiting | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  times /day.
Consistency of Vomiting | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Soft/ watery/ abnormal constitute
Duration of Vomiting | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  /days.
General condition of child | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Normal/ Restless, irritable/ Lethargic or unconscious
Eye | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Normal/ Sunken eyes/ Very Sunken eyes
Thirsty | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Drink normally/ Drinks eagerly, thirsty/ Drinks poorly or unable to drink
Skin pinch | before intervention, after 1st day of study, after 2nd day of study, and after 3rd day of study.
  Goes back quickly/ Goes back slowly/ Goes back very slowly

OTHER OUTCOMES:
children's age/ | before data collection
  year(s)
gender/ | before data collection
  male, female
residence/ | before data collection
  urban,rural
type of feeding | before data collection
  breast feeding, bottle feeding, mixed type, ordinary
diagnosis | before data collection
  gastroenteritis, bronchitis
prescribed medication | before data collection
  antiemetics, fluids therapy, antibiotics
children's weight | before data collection
  /kgs

CONTACTS AND LOCATIONS:
Locations (1):
- inpatient medical ward for gastroenteritis in El-Raml Children's Hospital (Wingat) at Alexandria., Alexandria, Egypt

REFERENCES:
- [Background] Bertelsen RJ, Jensen ET, Ringel-Kulka T. Use of probiotics and prebiotics in infant feeding. Best Pract Res Clin Gastroenterol. 2016 Feb;30(1):39-48. doi: 10.1016/j.bpg.2016.01.001. Epub 2016 Jan 22. PMID 27048895
- [Background] Cruchet S, Furnes R, Maruy A, Hebel E, Palacios J, Medina F, Ramirez N, Orsi M, Rondon L, Sdepanian V, Xochihua L, Ybarra M, Zablah RA. The use of probiotics in pediatric gastroenterology: a review of the literature and recommendations by Latin-American experts. Paediatr Drugs. 2015 Jun;17(3):199-216. doi: 10.1007/s40272-015-0124-6. PMID 25799959
- [Background] Kluijfhout S, Trieu TV, Vandenplas Y. Efficacy of the Probiotic Probiotical Confirmed in Acute Gastroenteritis. Pediatr Gastroenterol Hepatol Nutr. 2020 Sep;23(5):464-471. doi: 10.5223/pghn.2020.23.5.464. Epub 2020 Aug 27. PMID 32953642
- [Background] Sharif, A., Kheirkhah, D., Shamsesfandabadi, P., Masoudi, S., Ajorpaz, N., & Sharif, M. (2017, 01/01). Comparison of Regular and Probiotic Yogurts in Treatment of Acute Watery Diarrhea in Children. Journal of Probiotics & Health, 05. https://doi.org/10.4172/2329-8901.1000164